CLINICAL TRIAL: NCT00645788
Title: Randomized, Double-blind, Placebo-controlled, Multicenter Study to Evaluate the Safety and Efficacy of Inhaled Ciprofloxacin Compared to Placebo in Subjects With Cystic Fibrosis
Brief Title: Study to Evaluate the Safety and Efficacy of Ciprofloxacin (Inhaled) in Patients With Cystic Fibrosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 12429; 2008-008314-40 (EudraCT Number)
Record Dates: First submitted 2008-03-26; First posted 2008-03-28 (Estimated); Results first posted 2012-07-03 (Estimated); Last update posted 2014-06-09 (Estimated); Status verified 2014-05

CONDITIONS: Cystic Fibrosis
Keywords: Ciprofloxacin; cystic fibrosis; sweat test; pulmonary function test
MeSH Terms: conditions — Cystic Fibrosis | interventions — Ciprofloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 32.50 mg Ciprofloxacin DPI (BAYQ3939) (Experimental): 32.50 mg ciprofloxacin DPI (Dry Powder for Inhalation) corresponding to 50 mg Ciprofloxacin PulmoSphere Inhalation Powder twice a day for 28 days
  Interventions: Drug: Ciprofloxacin (Cipro Inhale, BAYQ3939)
- 48.75 mg Ciprofloxacin DPI (BAYQ3939) (Experimental): 48.75 mg ciprofloxacin DPI corresponding to 75 mg Ciprofloxacin PulmoSphere Inhalation Powder twice a day for 28 days
  Interventions: Drug: Ciprofloxacin (Cipro Inhale, BAYQ3939)
- Matching Placebo for 32.50 mg (Placebo Comparator): Inhalation of placebo powder formulation matching 32.50 mg ciprofloxacin DPI twice a day for 28 days
  Interventions: Drug: Placebo
- Matching Placebo for 48.75 mg (Placebo Comparator): Inhalation of placebo powder formulation matching 48.75 mg ciprofloxacin DPI twice a day for 28 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ciprofloxacin (Cipro Inhale, BAYQ3939) — 32.5 mg ciprofloxacin DPI corresponding to 50 mg Ciprofloxacin PulmoSphere Inhalation powder twice a day for 28 days
  Arms: 32.50 mg Ciprofloxacin DPI (BAYQ3939)
Drug: Placebo — 50 mg matching placebo powder formulation twice a day for 28 days
  Arms: Matching Placebo for 32.50 mg
Drug: Ciprofloxacin (Cipro Inhale, BAYQ3939) — 48.75 mg ciprofloxacin DPI corresponding to 75 mg Ciprofloxacin PulmoSphere Inhalation powder twice a day for 28 days (Arm 3 and Arm 4 was introduced after amendment 2)
  Arms: 48.75 mg Ciprofloxacin DPI (BAYQ3939)
Drug: Placebo — 75 mg matching placebo powder formulation twice a day for 28 days (Arm 3 and Arm 4 was introduced after amendment 2)
  Arms: Matching Placebo for 48.75 mg

SUMMARY:
To evaluate the change in forced expiratory volume (FEV1) from baseline to Day 28-30 between Cipro Inhale-treated and placebo-treated subjects after a 4-week treatment period.

DETAILED DESCRIPTION:
Safety issues are addressed in the Adverse Events section.

ELIGIBILITY:
Inclusion Criteria:

* Subjects, or their legal representative(s), must have given their written informed consent to participate in the study after receiving adequate previous information and prior to any study specific procedures
* Children (12 - 17 years) or adults >/=18 years
* Documented diagnosis Cystic Fibrosis (CF):

  * documented sweat chloride >/=60 mEq/L by quantitative pilocarpine iontophoresis test (QPIT) or nasal potential difference
  * either homozygous for ΔF508 genetic mutation or a compound heterozygous for 2 known CF mutations
  * and clinical findings consistent with CF
* Chronic colonization with P. aeruginosa defined as a positive respiratory tract culture (sputum or throat swab) within 12 months prior to screening and at screening (Note: subjects with negative culture at screening can, at the discretion of the investigator, be rescreened at a later date)
* Ability to perform reproducible pulmonary function tests
* Ability to produce sputum (noninduced)
* Stable pulmonary status, FEV1 >/=35% to </=75% (intraindividual variability +/-10% of absolute value). Note: The subject is not eligible for enrollment if the variability results in (or leads to) an FEV1 <35%.
* Room air oximetry >/=88% saturation
* Off antibiotics (except macrolide) and Cipro (oral) for at least 30 days prior to the administration of study drug for pulmonary exacerbation
* Stable regimen of standard CF treatment including chest physiotherapies and exercise regimens should not change during the 30 days prior to the administration of study drug and during the study (including macrolide administration unchanged in the previous 30 days)
* Subjects who are able to understand and follow instructions and who are able to participate in the study for the entire period
* Women who are willing to use an adequate method of contraception for 3 months after receiving the study drug. Adequate methods of contraception include vasectomy or condom use by their partners, diaphragm with spermicidal gel, coil (intrauterine device), surgical sterilization or oral contraceptive

Exclusion Criteria:

* Findings on screening history and physical examination unrelated to CF that could potentially affect the efficacy measurements (eg, chest surgery)
* Subjects with colonization of Pseudomonas aeruginosa and a CIPRO MIC of >/=256 µg/ml or mg/l
* Burkholderia cepacia complex colonization of their respiratory tract within the past 12 months (documented by screen laboratory)
* Known aspergillosis (unless asymptomatic). Patients with invasive disease, ABPA with IGE > 500 mg/dL will be excluded
* Transaminase level >3x upper limit of normal (ULN)
* Massive hemoptysis (>/=300 cc or requiring blood transfusion) in the preceding 4 weeks
* Intravenous antibiotic treatment for pulmonary exacerbation in the past 30 days
* Subjects with a medical disorder, condition or history of such that would impair the subject's ability to participate or complete this study in the opinion of the investigator or the sponsor
* Febrile illness within 1 week before the start of the study
* Active treatment for nontuberculosis mycobacteria
* Exposure to any investigational drug within 30 days
* Any history of allergic reaction to fluoroquinolones or other quinolones
* On oral steroids >20 mg/day for longer than 14 days in the past 3 months
* Creatinine >/=2x ULN

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 288 (Actual)
Dates: Start 2008-05; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (78):
- United States (50):
  - Phoenix, Arizona
  - Tucson, Arizona
  - Little Rock, Arkansas
  - Los Angeles, California
  - Orange, California
  - San Diego, California
  - San Francisco, California
  - Ventura, California
  - Aurora, Colorado
  - Hartford, Connecticut
  - New Haven, Connecticut
  - Jacksonville, Florida
  - Miami, Florida
  - Orlando, Florida
  - Augusta, Georgia
  - Chicago, Illinois
  - Glenview, Illinois
  - Maywood, Illinois
  - Indianapolis, Indiana
  - Iowa City, Iowa
  - Lexington, Kentucky
  - Louisville, Kentucky
  - Boston, Massachusetts
  - Ann Arbor, Michigan
  - Kalamazoo, Michigan
  - Jackson, Mississippi
  - Las Vegas, Nevada
  - Livingston, New Jersey
  - Long Branch, New Jersey
  - Morristown, New Jersey
  - Somerville, New Jersey
  - Albany, New York
  - New Hyde Park, New York
  - Valhalla, New York
  - Durham, North Carolina
  - Akron, Ohio
  - Cincinnati, Ohio
  - Toledo, Ohio
  - Oklahoma City, Oklahoma
  - Tulsa, Oklahoma
  - Hershey, Pennsylvania
  - Philadelphia, Pennsylvania
  - Charleston, South Carolina
  - Knoxville, Tennessee
  - Austin, Texas
  - San Antonio, Texas
  - Salt Lake City, Utah
  - Charlottesville, Virginia
  - Seattle, Washington
  - Madison, Wisconsin
- Australia (7):
  - Brisbane, Queensland
  - Chermside, Queensland
  - South Brisbane, Queensland
  - Adelaide, South Australia
  - Clayton, Victoria
  - Parkville, Victoria
  - Nedlands, Western Australia
- Canada (4):
  - St. John's, Newfoundland and Labrador
  - Hamilton, Ontario
  - London, Ontario
  - Montreal, Quebec
- Copenhagen, Denmark
- Germany (4):
  - München, Bavaria
  - Frankfurt am Main, Hesse
  - Leipzig, Saxony
  - Berlin, State of Berlin
- Israel (4):
  - Haifa
  - Jerusalem
  - Petah Tikva
  - Tel Litwinsky
- Oslo, Norway
- Sweden (3):
  - Gothenburg
  - Lund
  - Uppsala
- United Kingdom (4):
  - Cambridge, Cambridgeshire
  - Southampton, Hampshire
  - Belfast, North Ireland
  - Birmingham, West Midlands

REFERENCES:
- [Derived] Dorkin HL, Staab D, Operschall E, Alder J, Criollo M. Ciprofloxacin DPI: a randomised, placebo-controlled, phase IIb efficacy and safety study on cystic fibrosis. BMJ Open Respir Res. 2015 Dec 2;2(1):e000100. doi: 10.1136/bmjresp-2015-000100. eCollection 2015. PMID 26688732

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first visit of the first subject was on 05 May 2008 and the last visit of the last subject on 25 Jan 2011. This study was conducted at 73 centers from 8 countries.
Pre-assignment Details: Of all enrolled 486 subjects, 188 had screening failures, the remaining 288 were randomized but 2 subjects (one each in 32.5 mg Ciprofloxacin DPI (Dry Powder for Inhalation) and 48.75 mg Ciprofloxacin DPI groups) did not receive any study drug. A total of 286 subjects received one of the 4 study drug treatments.
Period: Overall Study
Arm/Group | 32.50 mg Ciprofloxacin DPI (BAYQ3939) | 48.75 mg Ciprofloxacin DPI (BAYQ3939) | Matching Placebo for 32.50 mg | Matching Placebo for 48.75 mg
Started | 94 | 94 | 65 | 35
Participants Receive Treatment | 93 | 93 | 65 | 35
Completed | 74 | 67 | 47 | 21
Not Completed | 20 | 27 | 18 | 14
Not completed — Did not receive study drug | 1 | 1 | 0 | 0
Not completed — Adverse Event | 4 | 9 | 5 | 3
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 2
Not completed — Pulmonary exacerbation | 13 | 16 | 11 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 32.50 mg Ciprofloxacin DPI (BAYQ3939) | 48.75 mg Ciprofloxacin DPI (BAYQ3939) | Matching Placebo for 32.50 mg | Matching Placebo for 48.75 mg | Total
Number analyzed (Participants) | 93 | 93 | 65 | 35 | 286
Age, Continuous [Mean (Standard Deviation); unit: Years] | 27.7 (9.3) | 29.3 (9.5) | 31.7 (12.1) | 29.1 (9.4) | 29.3 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 42 | 26 | 16 | 133
  Male | 44 | 51 | 39 | 19 | 153
Forced expiratory volume in 1 second (FEV1) [Mean (Standard Deviation); unit: Percentage of predicted FEV1] | 55.0 (11.3) | 54.7 (12.3) | 54.8 (10.6) | 52.7 (10.7) | 54.6 (11.4)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Forced Expiratory Volume in 1 Second (FEV1) at Day 28-30
Description: FEV1: The maximal volume of air exhaled in the first second of a forced expiration from a position of full inspiration, expressed in liters at body temperature and ambient pressure saturated with water vapor (BTPS). This was recorded at the site using a spirometer. The later time point minus baseline, days as planned and the last observation carried forward (LOCF) used.
Time Frame: Baseline and End of treatment (Day 28-30)
Population: Intent to treat
Measure: Mean (Standard Deviation); unit: Percent of predicted FEV1
Groups:
- 32.50 mg Ciprofloxacin DPI (BAYQ3939): 32.5 mg ciprofloxacin DPI (Dry Powder for Inhalation) corresponding to 50 mg Ciprofloxacin PulmoSphere Inhalation Powder twice a day for 28 days
Arm/Group | 32.50 mg Ciprofloxacin DPI (BAYQ3939) | 48.75 mg Ciprofloxacin DPI (BAYQ3939) | Matching Placebo for 32.50 mg | Matching Placebo for 48.75 mg
Number analyzed (Participants) | 93 | 93 | 65 | 35
Percent of predicted FEV1 | -1.0 (6.01) | -0.62 (5.52) | -2.2 (5.47) | -2.2 (5.17)
Statistical Analysis 1: Comparison: 32.50 mg Ciprofloxacin DPI (BAYQ3939) vs 48.75 mg Ciprofloxacin DPI (BAYQ3939) vs Matching Placebo for 32.50 mg vs Matching Placebo for 48.75 mg; Ho: |Cipro 32.5 mg - matching placebo|=0 and |Cipro 48.75 mg - matching placebo|=0; Test type: Superiority or Other; p = 0.076, ANCOVA

2. Secondary Outcome: Change From Baseline in FEV1 at Visits 4, 5, and Follow-up Visits 8 and 9
Description: as for outcome 1
Time Frame: Baseline and Visit 4 (Day 7-9), Visit 5 (Day 14-16), Visit 8 (Day 41-45), and Visit 9 (Day 56 -60).
Population: Intent to treat
Measure: Mean (Standard Deviation); unit: Percent of predicted FEV1
Arm/Group | 32.50 mg Ciprofloxacin DPI (BAYQ3939) | 48.75 mg Ciprofloxacin DPI (BAYQ3939) | Matching Placebo for 32.50 mg | Matching Placebo for 48.75 mg
Number analyzed (Participants) | 93 | 93 | 65 | 35
Percent of predicted FEV1
  Visit 4 | 0.40 (5.14) | 0.65 (4.62) | -0.84 (3.92) | -0.36 (3.5)
  Visit 5 | 0.10 (6.14) | 0.26 (3.94) | -1.6 (3.59) | -0.87 (4.00)
  Visit 8 | -1.5 (5.95) | -0.71 (5.14) | -1.2 (6.04) | -1.6 (5.23)
  Visit 9 | -2.0 (5.22) | -0.95 (5.29) | -1.9 (4.89) | -1.6 (5.13)

3. Secondary Outcome: Change From Baseline in P. Aeruginosa Density in the Sputum at Visits 4, 5, 7, 8 and 9
Description: Density of P. aeruginosa in the sputum is expressed as log10 of colony forming units (CFU)/gram (g). The later time point minus baseline, days as planned and the last observation carried forward (LOCF) used.
Time Frame: Baseline and Visit 4 (Day 7-9), Visit 5 (Day 14-16), Visit 7 (Day 28-30), Visit 8 (Day 41-45), and Visit 9 (Day 56 -60).
Population: Intent to treat
Measure: Mean (Standard Deviation); unit: log10(cfu/g)
Arm/Group | 32.50 mg Ciprofloxacin DPI (BAYQ3939) | 48.75 mg Ciprofloxacin DPI (BAYQ3939) | Matching Placebo for 32.50 mg | Matching Placebo for 48.75 mg
Number analyzed (Participants) | 93 | 93 | 65 | 35
log10(cfu/g)
  Visit 4 | -0.76 (2.21) | -1.1 (1.63) | -0.35 (2.09) | -0.56 (2.73)
  Visit 5 | -0.98 (2.51) | -1.0 (2.13) | 0.15 (2.06) | -0.65 (2.45)
  Visit 7 | -0.73 (2.57) | -0.78 (2.54) | -0.07 (2.59) | -0.63 (2.15)
  Visit 8 | -0.26 (2.52) | -0.11 (2.39) | -0.14 (2.21) | -0.00 (2.43)
  Visit 9 | 0.13 (2.19) | -0.16 (2.26) | -0.19 (2.15) | 0.54 (1.69)
Statistical Analysis 1: Comparison: 32.50 mg Ciprofloxacin DPI (BAYQ3939) vs 48.75 mg Ciprofloxacin DPI (BAYQ3939) vs Matching Placebo for 32.50 mg vs Matching Placebo for 48.75 mg; At visit 7 (End of treatment) Ho: |Cipro 32.5 - matching placebo| =0 and |Cipro 48.75 - matching placebo| =0; Test type: Superiority or Other; p = 0.068, ANCOVA

4. Secondary Outcome: Time to First Pulmonary Exacerbation Requiring Intervention
Description: Pulmonary exacerbations: Assessment of pulmonary exacerbation was conducted by the treating physician as part of the physical examination. Pulmonary exacerbation was defined by chest examination findings and any or all of the following symptoms: decreased exercise tolerance, increased cough, increased sputum/cough congestion, school or work absenteeism, increased adventitial sounds on the lung examination, and decreased appetite.
Time Frame: Up to visit 9 (Day 56-60)
Population: Intent to treat
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | 32.50 mg Ciprofloxacin DPI (BAYQ3939) | 48.75 mg Ciprofloxacin DPI (BAYQ3939) | Matching Placebo for 32.50 mg | Matching Placebo for 48.75 mg
Number analyzed (Participants) | 93 | 93 | 65 | 35
Days | NA [NA to NA] — only 16.1 percent of patients had an exacerbation | NA [NA to NA] — only 17.2 percent of patients had an exacerbation | NA [NA to NA] — only 20.0 percent of patients had an exacerbation | NA [43 to NA] — only 28.6 percent of patients had an exacerbation

5. Secondary Outcome: Change From Baseline in Forced Vital Capacity (FVC) at Visits 4, 5, 7, 8 and 9
Description: FVC: The maximal volume of air exhaled with maximally forced effort from a maximal inspiration, ie, vital capacity performed with a maximally forced expiratory effort expressed in liters at BTPS (body temperature and ambient pressure saturated with water vapor). The later time point minus baseline, days as planned and the last observation carried forward (LOCF) used.
Time Frame: Baseline and Visit 4 (Day 7-9), Visit 5 (Day 14-16), Visit 7 (Day 28-30), Visit 8 (Day 41-45), and Visit 9 (Day 56 -60).
Population: Intent to treat
Measure: Mean (Standard Deviation); unit: Percent of predicted FVC
Arm/Group | 32.50 mg Ciprofloxacin DPI (BAYQ3939) | 48.75 mg Ciprofloxacin DPI (BAYQ3939) | Matching Placebo for 32.50 mg | Matching Placebo for 48.75 mg
Number analyzed (Participants) | 93 | 93 | 65 | 35
Percent of predicted FVC
  Visit 4 | -2.5 (8.97) | 0.22 (5.07) | -0.94 (5.23) | -0.45 (4.98)
  Visit 5 | -2.2 (9.78) | -0.48 (5.11) | -1.8 (4.51) | -1.1 (5.57)
  Visit 7 | -2.8 (8.91) | -1.4 (6.04) | -2.7 (6.97) | -1.4 (8.41)
  Visit 8 | -2.6 (8.62) | -0.65 (6.44) | -1.6 (7.31) | 0.13 (7.72)
  Visit 9 | -2.9 (8.54) | -0.70 (6.64) | -2.3 (5.63) | -0.53 (7.37)

6. Secondary Outcome: Change From Baseline in Forced Expiratory Flow (FEF 25-75%) at Visits 4, 5, 7, 8 and 9
Description: FEF 25-75% (also known as the maximum midexpiratory flow [MMEF]): The mean forced expiration flow over the middle half of the forced vital capacity (FVC). It was taken from the blow with the largest sum of FEV1 and FVC. The later time point minus baseline, days as planned and the last observation carried forward (LOCF) used.
Time Frame: Baseline and Visit 4 (Day 7-9), Visit 5 (Day 14-16), Visit 7 (Day 28-30), Visit 8 (Day 41-45), and Visit 9 (Day 56 -60).
Population: Intent to treat
Measure: Mean (Standard Deviation); unit: Percent of predicted FEF 25-75%
Arm/Group | 32.50 mg Ciprofloxacin DPI (BAYQ3939) | 48.75 mg Ciprofloxacin DPI (BAYQ3939) | Matching Placebo for 32.50 mg | Matching Placebo for 48.75 mg
Number analyzed (Participants) | 93 | 93 | 65 | 35
Percent of predicted FEF 25-75%
  Visit 4 | 2.13 (7.12) | 1.09 (6.90) | -1.0 (4.65) | -0.49 (4.55)
  Visit 5 | 1.48 (8.16) | 0.95 (4.73) | -1.1 (4.49) | -0.89 (4.16)
  Visit 7 | 0.24 (6.84) | 0.35 (5.39) | -2.1 (5.62) | -1.8 (4.73)
  Visit 8 | 0.16 (7.56) | -0.33 (5.19) | -1.2 (6.23) | -1.9 (5.31)
  Visit 9 | -0.46 (7.35) | -0.49 (5.55) | -1.3 (5.63) | -1.4 (4.99)

7. Secondary Outcome: Number of Participants Developing Ciprofloxacin-resistant Mucoid P.Aeruginosa Isolates
Description: Susceptibility and resistance assessment of a bacterial isolate was performed using the established Food and Drug Administration (FDA) susceptibility criteria for ciprofloxacin. The susceptibility criteria in mg/L are ≤1 for organisms Enterobacteriaciae, P. aeruginosa, Staphylococcus species and S. pneumoniae. The "susceptible" bacterial species likely responds to typical doses of ciprofloxacin. The resistance criteria for ciprofloxacin in mg/L are ≥4 mg/L for the same organisms. Resistance indicates that the bacteria is less likely to respond to typical doses of ciprofloxacin therapy.
Time Frame: Baseline and up to visit 9 (day 56-60)
Population: Intent to treat
Measure: Number; unit: Participants
Arm/Group | 32.50 mg Ciprofloxacin DPI (BAYQ3939) | 48.75 mg Ciprofloxacin DPI (BAYQ3939) | Matching Placebo for 32.50 mg | Matching Placebo for 48.75 mg
Number analyzed (Participants) | 93 | 93 | 65 | 35
Participants
  P.aeruginosa sensitive - baseline | 70 | 60 | 51 | 30
  P.aeruginosa resistant - up to visit 9 | 15 | 15 | 11 | 3

8. Secondary Outcome: Number of Participants Developing Ciprofloxacin-resistant Non-mucoid P.Aeruginosa Isolates
Description: as for outcome 7
Time Frame: Baseline and up to visit 9 (day 56-60)
Population: Intent to treat
Measure: Number; unit: Participants
Arm/Group | 32.50 mg Ciprofloxacin DPI (BAYQ3939) | 48.75 mg Ciprofloxacin DPI (BAYQ3939) | Matching Placebo for 32.50 mg | Matching Placebo for 48.75 mg
Number analyzed (Participants) | 93 | 93 | 65 | 35
Participants
  P.aeruginosa sensitive - baseline | 72 | 63 | 48 | 23
  P.aeruginosa resistant- up to visit 9 | 29 | 31 | 19 | 7

9. Secondary Outcome: Effect of Ciprofloxacin DPI Treatment on Quality of Life Measured by Cystic Fibrosis Quality of Life Questionnaire Revised (CFQ-R), Respiratory Scale
Description: The CF quality of life questionnaire revised (CFQ-R), a validated disease-specific instrument that measures health-related quality of life (HRQOL) for adolescents and adults with cystic fibrosis (CF). It is self-administered and consists of 44 items, divided into 12 generic and disease-specific scales. The scale includes physical functioning, role, vitality, emotional functioning, social functioning, body image, eating disturbances, treatment burden, health perceptions, weight, respiratory symptoms, and digestive symptoms. Scale range: 0 to 100 (maximum). Better outcome with higher values.
Time Frame: Baseline and Visit 7 (Day 28-30) and Visit 9 (Day 56 -60)
Population: Intent to treat
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | 32.50 mg Ciprofloxacin DPI (BAYQ3939) | 48.75 mg Ciprofloxacin DPI (BAYQ3939) | Matching Placebo for 32.50 mg | Matching Placebo for 48.75 mg
Number analyzed (Participants) | 93 | 93 | 65 | 35
scores on a scale
  Baseline | 68.0 (18.7) | 59.5 (19.0) | 61.3 (18.6) | 68.3 (13.8)
  Visit 7 | 70.8 (15.9) | 60.0 (19.7) | 58.9 (18.7) | 61.6 (18.4)
  Visit 9 | 67.2 (18.9) | 60.6 (20.5) | 61.1 (19.8) | 71.2 (16.6)

10. Secondary Outcome: Plasma Concentrations of Ciprofloxacin From Selected Participants During Treatment
Description: Plasma concentrations measured using validated high pressure liquid chromatography-mass specroscopy/mass spectroscopy (HPLC-MS/MS) methods in selected patients at predefined time windows to contribute pharmacokinetic (PK) information for an inter-study population PK evaluation. Sampling window for Plasma: Predose (trough level), <15 min, 2.0 - 2.5 hour, and 4.0 - 7.0 hours after the end of inhalation. Number of samples vary at different time points.
Time Frame: Up to visit 7 (Day 28-30)
Population: Analysis was not performed due to insufficient data.
Arm/Group | 32.50 mg Ciprofloxacin DPI (BAYQ3939) | 48.75 mg Ciprofloxacin DPI (BAYQ3939)
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Sputum Concentrations of Ciprofloxacin From Selected Participants During Treatment
Description: Sputum concentrations measured using validated HPLC-MS/MS methods in selected patients to contribute kinetic information for an inter-study population sputum kinetic evaluation. Number of samples vary at different time points.
Time Frame: Up to visit 7 (Day 28-30)
Population: Analysis was not performed due to insufficient data.
Arm/Group | 32.50 mg Ciprofloxacin DPI (BAYQ3939) | 48.75 mg Ciprofloxacin DPI (BAYQ3939)
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Number of Participants With the Occurrence of Drug Induced Bronchospasms
Description: Bronchospasm reported as adverse event: Bronchospasm defined as >=15% drop in FEV1, and may also include allergic and excercise-induced bronchospasm. Drug-induced bronchospasm: Treatment-emergent bronchospasm was defined as >=15% drop in FEV1 in the ITT/safety population. Note: One of the bronchospasm events was considered a serious adverse event, and it was not included under "other" adverse events. A sum of bronchospasm events was 1+6=7.
Time Frame: Up to visit 9 (Day 56-60)
Population: Intent to treat
Measure: Number; unit: participants
Arm/Group | 32.50 mg Ciprofloxacin DPI (BAYQ3939) | 48.75 mg Ciprofloxacin DPI (BAYQ3939) | Matching Placebo for 32.50 mg | Matching Placebo for 48.75 mg
Number analyzed (Participants) | 93 | 93 | 65 | 35
participants
  Reported as Adverse event | 4 | 7 | 3 | 0
  Defined as >=15 percent drop in FEV1 | 3 | 3 | 3 | 0

ADVERSE EVENTS:
Arm/Group | 32.50 mg Ciprofloxacin DPI (BAYQ3939) | 48.75 mg Ciprofloxacin DPI (BAYQ3939) | Matching Placebo for 32.50 mg | Matching Placebo for 48.75 mg
Serious Adverse Events (participants affected / at risk) | 7/93 | 17/93 | 7/65 | 3/35
Other Adverse Events (participants affected / at risk) | 67/93 | 74/93 | 45/65 | 25/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 32.50 mg Ciprofloxacin DPI (BAYQ3939) (N=93) | 48.75 mg Ciprofloxacin DPI (BAYQ3939) (N=93) | Matching Placebo for 32.50 mg (N=65) | Matching Placebo for 48.75 mg (N=35)
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Distal intestinal obstruction syndrome (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Bronchopneumonia (Infections and infestations) | 0 | 0 | 1 | 0
H1N1 influenza (Infections and infestations) | 1 | 0 | 0 | 0
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 5 | 11 | 4 | 3
Sinusitis (Infections and infestations) | 0 | 0 | 1 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 32.50 mg Ciprofloxacin DPI (BAYQ3939) (N=93) | 48.75 mg Ciprofloxacin DPI (BAYQ3939) (N=93) | Matching Placebo for 32.50 mg (N=65) | Matching Placebo for 48.75 mg (N=35)
Nausea (Gastrointestinal disorders) | 2 | 4 | 1 | 2
Chest discomfort (General disorders) | 5 | 4 | 5 | 0
Exercise tolerance decreased (General disorders) | 2 | 4 | 1 | 2
Product taste abnormal (General disorders) | 7 | 16 | 4 | 2
Pyrexia (General disorders) | 2 | 2 | 4 | 0
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 22 | 18 | 10 | 11
Nasopharyngitis (Infections and infestations) | 1 | 6 | 0 | 2
Upper respiratory tract infection (Infections and infestations) | 4 | 8 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 5 | 5 | 3 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 2 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 5 | 0 | 0
Dysgeusia (Nervous system disorders) | 13 | 9 | 4 | 1
Headache (Nervous system disorders) | 1 | 4 | 7 | 2
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 4 | 6 | 3 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 24 | 20 | 22 | 10
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 | 3 | 2 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 7 | 7 | 5 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 5 | 2 | 4 | 1
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 4 | 7 | 1 | 0
Rales (Respiratory, thoracic and mediastinal disorders) | 8 | 8 | 2 | 2
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 5 | 3 | 3 | 1
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 5 | 3 | 0 | 2
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 12 | 11 | 11 | 5
Wheezing (Respiratory, thoracic and mediastinal disorders) | 5 | 7 | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The agreed point of publication is 12-18 months after database lock at the earliest. Bayer will have 30-45 days to review publications, and may request an additional publication delay of up to 60 days to allow for filing a Patent Application (if applicable). No publication of single center data should be done prior of publication if multi-center data.